CLINICAL TRIAL: NCT04870723
Title: An International Multi-site, Randomized Controlled Trial of a Brief eHealth Intervention to Increase COVID-19 Knowledge and Protective Behaviors, and Reduce Pandemic Stress Among Diverse LGBT+ People
Brief Title: #SafeHandsSafeHearts: An eHealth Intervention for COVID-19 Prevention and Support
Acronym: COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Responsible Party: Principal Investigator, Peter A. Newman, Professor, University of Toronto
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 39769
Record Dates: First submitted 2021-04-23; First posted 2021-05-03 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Covid19
Keywords: COVID-19; Protective behaviors; LGBT populations; Racialized populations; Social determinants of health; Randomized controlled trial; Psychoeducation; Motivational-interviewing; Low- and middle-income countries; Psychological distress
MeSH Terms: conditions — COVID-19 | interventions — Telemedicine; Palliative Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate (Experimental): Behavioral: Motivational interviewing (MI)-based peer counseling: MI-based peer counseling will comprise of 3 weekly 1-hour sessions administered online addressing 1) Covid-19 knowledge; 2) Assessing risk for infection and understanding and practicing public health-recommended protective behaviors (masking, physical distancing, handwashing); and 3) Understanding psychosocial issues and maintaining mental wellness.
  Interventions: Behavioral: eHealth for Covid-19 prevention and support
- Waitlist (Other): Behavioral: Motivational interviewing (MI)-based peer counseling: After the immediate group completes the intervention, the waitlist group will receive the intervention.
  MI-based peer counseling will comprise of 3 weekly 1-hour sessions administered online addressing 1) Covid-19 knowledge; 2) Assessing risk for infection and understanding and practicing public health-recommended protective behaviors (masking, physical distancing, handwashing); and 3) Understanding psychosocial issues and maintaining mental wellness.
  Interventions: Behavioral: eHealth for Covid-19 prevention and support

INTERVENTIONS:
Behavioral: eHealth for Covid-19 prevention and support — 3-session online peer-counseling intervention based on motivational interviewing and psychoeducation

SUMMARY:
This project seeks to test the efficacy of a brief eHealth intervention in an international randomized controlled trial (RCT) to increase COVID-19 knowledge and protective behaviors, and reduce psychological distress among LGBT people. This project involves enrolling racially diverse samples of lesbian, gay, bisexual and transgender people in three cities, randomizing 900 people (stratified among cisengender men, cisgender women, and transgender people) to either the immediate behavioral intervention or the waitlist control condition. Participants will complete a baseline survey, a follow-up survey 2 weeks post-intervention, and a final survey 2 months after the post-intervention survey. Primary outcomes are COVID-19 transmission knowledge, COVID-19 protective behaviors, and psychological distress.

DETAILED DESCRIPTION:
Lesbian, gay, bisexual, and transgender (LGBT+) populations are at heightened vulnerability to COVID-19 due to existing health disparities amid adverse social determinants of health (SDOH), rights violations, and social-structural constraints on public health recommended (PHR) protective measures. Yet, public health responses largely do not address LGBT+ vulnerabilities nor do they include LGBT+ communities in pandemic response planning.

As there is no manualized intervention for COVID-19 prevention, the investigators will adapt an efficacious eHealth intervention for preventing HIV infection and transmission, the deadliest pandemic of the last century. This study builds on evidence-based eHealth interventions using Motivational Interviewing (MI) and Psychoeducation to increase health knowledge and behaviors, and reduce psychological distress, including interventions with LGBT+ people.

MI is a client-centered counseling approach that elicits and strengthens intrinsic motivation for change. Psychoeducation integrates education and counseling to promote mental health. Peer counselors will receive 5 days of online training on COVID-19, PHR behaviors, pandemic stress (anxiety, depression, social isolation), MI-based counselling, psychoeducation, and research ethics. The 3 primary study outcomes are increasing COVID-19 knowledge, PHR protective behaviors, and reducing psychological distress; these are crucial elements of public health approaches to control SARS-CoV-2 transmission.

#SafeHandsSafeHearts is a 3-session peer-delivered MI-based brief counselling (45 min-1 hr) with weekly individual sessions. Participants will be recruited online with electronic flyers and social media messages developed with community-based organization (CBO) partners, and distributed through CBO social media accounts and listservs in each of the three study sites (Toronto, Bangkok, Mumbai), and a study website. Participants will be randomized to the immediate intervention group or waitlist control group at a 1:1 ratio, stratified by sex and gender (cisgender men, cisgender women, transgender people), using a computer-generated sequence. All participants will complete a baseline survey, a post-intervention follow-up survey 2 weeks after completing the intervention, and a final survey 2 months after post-intervention survey.

NOTE: Due to pandemic-related delays and lockdowns, and Toronto site ethics approvals and opening 6+ months prior to Bangkok and Mumbai sites, the Toronto site was conducted as a pilot intervention, using a pre-test post-test quasi-experimental design, to inform feasibility, acceptability, and implementation of the eHealth intervention, and provide initial outcomes. Bangkok and Mumbai sites remained RCTs. All sites used the prospectively identified study procedures including enrollment criteria, eHealth intervention, and baseline, post-intervention, and 2-month follow-up assessments.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Self-identified as LGBT+
* Lived in the study locale (city/region) for at least 6 months
* Plan to remain in the study locale (city/region) for at least 3 months

Exclusion Criteria:

* Located outside of Greater Toronto and Hamilton Area (Canada), Mumbai/Thane (India) or Bangkok metropolitan area (Thailand)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Self-identified as LGBT+
Enrollment: 853 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-05-15 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Change in COVID-19 knowledge | Baseline survey, 2-week post-intervention survey, and 2-month post-intervention survey
  COVID-19 transmission knowledge (index of 8 items, minimum score = 0 - maximum score = 8, higher score = greater knowledge/better outcome, based on CDC, 2020 [June 30])
Change in COVID-19 protective behaviors | Baseline survey, 2-week post-intervention survey, and 2-month post-intervention survey
  Mask wearing, physical distancing, handwashing (index of 9 items, minimum score = 0 - maximum score = 18, higher score = better outcome; based on CDC, 2020 [July 31])
Change in depressive symptoms | Baseline survey, 2-week post-intervention survey, and 2-month post-intervention survey
  Frequency of depressed mood and anhedonia (Patient Health Questionnaire 2 [PHQ-2], minimum score = 0, maximum score = 6; higher score = worse outcome)
Change in anxiety symptoms | Baseline survey, 2-week post-intervention survey, and 2-month post-intervention survey
  Frequency of anxiety symptoms (Generalized Anxiety Disorder 2 [GAD-2], minimum score = 0, maximum score = 6; higher score = worse outcome)

SECONDARY OUTCOMES:
Change in loneliness/social isolation | Baseline survey, 2-week post-intervention survey, and 2-month post-intervention survey
  Frequency of feeling lonely/socially isolated (Three-Item Loneliness Scale, minimum score = 0, maximum score = 6; higher score = worse outcome)

CONTACTS AND LOCATIONS:
Locations (3):
- Women's Health in Women's Hands, Toronto, Ontario, Canada
- Humsafar Trust, Mumbai, Maharashtra, India
- Institute of HIV Research and Innovation, Bangkok, Thailand

REFERENCES:
- [Background] Bandura, A. (1986). Social foundations of thought and action: A social cognitive theory. Prentice-Hall.
- [Background] Berg RC, Ross MW, Tikkanen R. The effectiveness of MI4MSM: how useful is motivational interviewing as an HIV risk prevention program for men who have sex with men? A systematic review. AIDS Educ Prev. 2011 Dec;23(6):533-49. doi: 10.1521/aeap.2011.23.6.533. PMID 22201237
- [Background] Betsch C. How behavioural science data helps mitigate the COVID-19 crisis. Nat Hum Behav. 2020 May;4(5):438. doi: 10.1038/s41562-020-0866-1. PMID 32221514
- [Background] Canadian Institutes of Health Research (CIHR). (2020). Why sex and gender need to be considered in COVID-19 research. https://cihr-irsc.gc.ca/e/51939.html
- [Background] Chakrapani V, Kaur M, Tsai AC, Newman PA, Kumar R. The impact of a syndemic theory-based intervention on HIV transmission risk behaviour among men who have sex with men in India: Pretest-posttest non-equivalent comparison group trial. Soc Sci Med. 2022 Feb;295:112817. doi: 10.1016/j.socscimed.2020.112817. Epub 2020 Jan 27. PMID 32033868
- [Background] Chiasson MA, Shaw FS, Humberstone M, Hirshfield S, Hartel D. Increased HIV disclosure three months after an online video intervention for men who have sex with men (MSM). AIDS Care. 2009 Sep;21(9):1081-9. doi: 10.1080/09540120902730013. PMID 20024766
- [Background] DiClemente CC, Corno CM, Graydon MM, Wiprovnick AE, Knoblach DJ. Motivational interviewing, enhancement, and brief interventions over the last decade: A review of reviews of efficacy and effectiveness. Psychol Addict Behav. 2017 Dec;31(8):862-887. doi: 10.1037/adb0000318. PMID 29199843
- [Background] Donker T, Griffiths KM, Cuijpers P, Christensen H. Psychoeducation for depression, anxiety and psychological distress: a meta-analysis. BMC Med. 2009 Dec 16;7:79. doi: 10.1186/1741-7015-7-79. PMID 20015347
- [Background] Eaton LA, Kalichman SC. Social and behavioral health responses to COVID-19: lessons learned from four decades of an HIV pandemic. J Behav Med. 2020 Jun;43(3):341-345. doi: 10.1007/s10865-020-00157-y. Epub 2020 Apr 25. PMID 32333185
- [Background] Frost H, Campbell P, Maxwell M, O'Carroll RE, Dombrowski SU, Williams B, Cheyne H, Coles E, Pollock A. Effectiveness of Motivational Interviewing on adult behaviour change in health and social care settings: A systematic review of reviews. PLoS One. 2018 Oct 18;13(10):e0204890. doi: 10.1371/journal.pone.0204890. eCollection 2018. PMID 30335780
- [Background] Gorgos LM, Marrazzo JM. Sexually transmitted infections among women who have sex with women. Clin Infect Dis. 2011 Dec;53 Suppl 3:S84-91. doi: 10.1093/cid/cir697. PMID 22080273
- [Background] Guse K, Levine D, Martins S, Lira A, Gaarde J, Westmorland W, Gilliam M. Interventions using new digital media to improve adolescent sexual health: a systematic review. J Adolesc Health. 2012 Dec;51(6):535-43. doi: 10.1016/j.jadohealth.2012.03.014. Epub 2012 May 5. PMID 23174462
- [Background] Hart TA, Stratton N, Coleman TA, Wilson HA, Simpson SH, Julien RE, Hoe D, Leahy B, Maxwell J, Adam BD. A Pilot Trial of a Sexual Health Counseling Intervention for HIV-Positive Gay and Bisexual Men Who Report Anal Sex without Condoms. PLoS One. 2016 Apr 7;11(4):e0152762. doi: 10.1371/journal.pone.0152762. eCollection 2016. PMID 27054341
- [Background] Hatzenbuehler ML, Phelan JC, Link BG. Stigma as a fundamental cause of population health inequalities. Am J Public Health. 2013 May;103(5):813-21. doi: 10.2105/AJPH.2012.301069. Epub 2013 Mar 14. PMID 23488505
- [Background] Herbst JH, Sherba RT, Crepaz N, Deluca JB, Zohrabyan L, Stall RD, Lyles CM; HIV/AIDS Prevention Research Synthesis Team. A meta-analytic review of HIV behavioral interventions for reducing sexual risk behavior of men who have sex with men. J Acquir Immune Defic Syndr. 2005 Jun 1;39(2):228-41. PMID 15905741
- [Background] Heslin KC, Hall JE. Sexual Orientation Disparities in Risk Factors for Adverse COVID-19-Related Outcomes, by Race/Ethnicity - Behavioral Risk Factor Surveillance System, United States, 2017-2019. MMWR Morb Mortal Wkly Rep. 2021 Feb 5;70(5):149-154. doi: 10.15585/mmwr.mm7005a1. PMID 33539330
- [Background] Higa DH, Crepaz N, Marshall KJ, Kay L, Vosburgh HW, Spikes P, Lyles CM, Purcell DW. A systematic review to identify challenges of demonstrating efficacy of HIV behavioral interventions for gay, bisexual, and other men who have sex with men (MSM). AIDS Behav. 2013 May;17(4):1231-44. doi: 10.1007/s10461-013-0418-z. PMID 23397183
- [Background] Lukens, E. P., & McFarlane, W. R. (2004). Psychoeducation as evidence-based practice: Considerations for practice, research, and policy. Brief Treatment and Crisis Intervention, 4(1), 205-25. https://doi.org/10.1093/brief-treatment/mhh019
- [Background] Markland, D., Ryan, R. M., Tobin V. J., Rollnick, S. (2005). Motivational interviewing and self-determination theory. Journal of Social and Clinical Psychology, 24(6), 811-311. https://doi.org/10.1521/jscp.2005.24.6.811
- [Background] Miller WR, Rollnick S. Meeting in the middle: motivational interviewing and self-determination theory. Int J Behav Nutr Phys Act. 2012 Mar 2;9:25. doi: 10.1186/1479-5868-9-25. No abstract available. PMID 22385872
- [Background] Miller, W.R., & Rollnick, S. (2002). Motivational interviewing: preparing people for change (2nd ed). Guilford Press.
- [Background] Naar-King S, Parsons JT, Johnson AM. Motivational interviewing targeting risk reduction for people with HIV: a systematic review. Curr HIV/AIDS Rep. 2012 Dec;9(4):335-43. doi: 10.1007/s11904-012-0132-x. PMID 22890780
- [Background] National Statistical Office and United Nations Children's Fund. (2016). Thailand multiple indicator cluster survey 2015-2016, final report. NSO and UNICEF, Thailand.
- [Background] Patel VV, Rawat S, Dange A, Lelutiu-Weinberger C, Golub SA. An Internet-Based, Peer-Delivered Messaging Intervention for HIV Testing and Condom Use Among Men Who Have Sex With Men in India (CHALO!): Pilot Randomized Comparative Trial. JMIR Public Health Surveill. 2020 Apr 16;6(2):e16494. doi: 10.2196/16494. PMID 32297875
- [Background] Prokopenko, E, & Kevins, C. (2020). Vulnerabilities related to COVID-19 among LGBTQ2+ Canadians. Statistic Canada. https://www150.statcan.gc.ca/n1/pub/45-28-0001/2020001/article/00075-eng.htm
- [Background] Razai MS, Osama T, McKechnie DGJ, Majeed A. Covid-19 vaccine hesitancy among ethnic minority groups. BMJ. 2021 Feb 26;372:n513. doi: 10.1136/bmj.n513. No abstract available. PMID 33637577
- [Background] Smedslund G, Berg RC, Hammerstrom KT, Steiro A, Leiknes KA, Dahl HM, Karlsen K. Motivational interviewing for substance abuse. Cochrane Database Syst Rev. 2011 May 11;2011(5):CD008063. doi: 10.1002/14651858.CD008063.pub2. PMID 21563163
- [Background] van Daalen KR, Bajnoczki C, Chowdhury M, Dada S, Khorsand P, Socha A, Lal A, Jung L, Alqodmani L, Torres I, Ouedraogo S, Mahmud AJ, Dhatt R, Phelan A, Rajan D. Symptoms of a broken system: the gender gaps in COVID-19 decision-making. BMJ Glob Health. 2020 Oct;5(10):e003549. doi: 10.1136/bmjgh-2020-003549. No abstract available. PMID 33004348
- [Derived] Newman PA, Chakrapani V, Massaquoi N, Williams CC, Tharao W, Tepjan S, Roungprakhon S, Forbes J, Sebastian S, Akkakanjanasupar P, Aden M. Effectiveness of an eHealth intervention for reducing psychological distress and increasing COVID-19 knowledge and protective behaviors among racialized sexual and gender minority adults: A quasi-experimental study (#SafeHandsSafeHearts). PLoS One. 2024 May 3;19(5):e0280710. doi: 10.1371/journal.pone.0280710. eCollection 2024. PMID 38701074
- [Derived] Newman PA, Chakrapani V, Williams C, Massaquoi N, Tepjan S, Roungprakhon S, Akkakanjanasupar P, Logie C, Rawat S. An eHealth Intervention for Promoting COVID-19 Knowledge and Protective Behaviors and Reducing Pandemic Distress Among Sexual and Gender Minorities: Protocol for a Randomized Controlled Trial (#SafeHandsSafeHearts). JMIR Res Protoc. 2021 Dec 10;10(12):e34381. doi: 10.2196/34381. PMID 34726610